CLINICAL TRIAL: NCT01661764
Title: Fatty Acid Desaturase Activity, Fish Oil and Colorectal Cancer Prevention
Brief Title: Fish Oil Supplementation, Nutrigenomics and Colorectal Cancer Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Harvey Murff, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11165; R01CA160938 (NIH)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Adenomatous Polyps
Keywords: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Eicosapentaenoic Acid; Omacor; Oleic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- rs174535 (GG), fish oil supplements (Active Comparator): Eicosapentanoic acid and docosahexanoic acid
  Interventions: Drug: Eicosapentanoic acid and docosahexanoic acid
- rs174535 (GG), placebo (Placebo Comparator): Oleic Acid
  Interventions: Drug: Oleic Acid
- rs174535 (GT), fish oil supplements (Active Comparator): Eicosapentanoic acid and docosahexanoic acid
  Interventions: Drug: Eicosapentanoic acid and docosahexanoic acid
- rs174535 (GT), placebo (Placebo Comparator): Oleic Acid
  Interventions: Drug: Oleic Acid
- rs174535 (TT), fish oil supplement (Active Comparator): Eicosapentanoic acid and docosahexanoic acid
  Interventions: Drug: Eicosapentanoic acid and docosahexanoic acid
- rs174535 (TT), placebo (Placebo Comparator): Oleic Acid
  Interventions: Drug: Oleic Acid

INTERVENTIONS:
Drug: Eicosapentanoic acid and docosahexanoic acid — 1395 mg EPA plus 1125 mg DHA daily for 24 weeks
  Other Names: Lovaza
  Arms: rs174535 (GG), fish oil supplements; rs174535 (GT), fish oil supplements; rs174535 (TT), fish oil supplement
Drug: Oleic Acid — Placebo
  Arms: rs174535 (GG), placebo; rs174535 (GT), placebo; rs174535 (TT), placebo

SUMMARY:
Colorectal cancer is the second leading cause of cancer-related death within the United States. Animal models and observational studies have suggested that marine-derived n-3 polyunsaturated fatty acids [PUFA] such as eicosapentanoic acid [EPA] and docosahexanoic acid [DHA] may reduce the risk of colorectal cancer. In addition, it may be the relative proportion of n-3 to n-6 PUFAs that best determines the chemopreventive effects of fish oils. This ratio is important because the n-6 PUFA, arachidonic acid (ARA), is converted via the cyclo-oxygenase (COX) pathway to prostaglandin E2 (PGE2), an inflammatory eicosanoid overproduced in colorectal neoplasms while EPA is converted to the anti-inflammatory prostaglandin E3 (PGE3). While the ratio of n-6 to n-3 PUFAs can be altered through dietary changes, genetic factors may also influence this ratio. Recent genetic studies have demonstrated that much of the tissue levels of ARA is determined by differences in a gene called fatty acid desaturase 1 (FADS1). FADS1 is the rate-limiting enzyme in the conversion of linoleic acid, the most commonly consumed PUFA in the Western diet, to ARA, and one particular genetic variant caller rs174537 is associated with lower fatty acid desaturase activity and subsequently lower tissue levels of ARA.

The study hypothesis is that individuals with genetically determined lower activity of FADS1 will derive greater benefit from fish oil supplementation than individuals with higher FADS1 activity because of lower tissue levels of ARA and subsequently a more favorable n-6 to n-3 PUFA ratio. To test this hypothesis the investigators will recruit 150 participants with recently identified adenomatous polyps and conduct a 6-month double blind 3 X 2 factorial randomized controlled trial. The first factor will be FADS1 genotype (GG, GT, and TT) and the second factor will be fish oil supplementation (fish oil versus placebo). The primary outcome will be the change in rectal epithelial cell growth and cell death. Secondary outcomes will include rectal epithelial cell expression of genes important in PGE2 production, rectal cell production of PGE2 and PGE3, rectal mucosal tissue levels of fatty acids, and changes in biomarkers of inflammation (C-reactive protein), adipokines (leptin, adiponectin), and markers of insulin sensitivity.

The specific aims include: 1) to determine the efficacy of fish oil supplements on rectal epithelial cell proliferation indexes and markers of rectal crypt apoptosis, and 2) to determine the effect of genetically-determined fatty acid desaturase 1 activity on fish oil supplementation for colorectal cancer chemoprevention. The investigators long-term objectives are to determine genetic factors that might influence the efficacy of fish oil supplementation in order to conduct a more definitive adenoma recurrence trial using marine-derived n-3 PUFAs. The investigators anticipate that fish oil will have anti-neoplastic effect and individuals with low FADS1 activity will have a greater response compared to individuals with high FADS1 activity

DETAILED DESCRIPTION:
1.Rationale and Specific Aims

Colorectal cancer (CRC) is the third most common cancer and the second most frequent cause of cancer related mortality in the United States. Animal and human studies have suggested that the marine-derived n-3 polyunsaturated fatty acids (PUFAs), eicosapentanoic acid (EPA) and docosahexanoic acid (DHA), have cancer inhibitory properties while conversely, n-6 PUFAs such as arachidonic acid (ARA) may promote tumorigenesis. The mechanism behind these opposing effects is likely due to differences in the biological activity of their eicosanoids end products and their effects on chronic inflammation. Prostaglandin E2 (PGE2) is a pro-inflammatory eicosanoid that is aberrantly produced in both colorectal adenomas and cancer and is derived from ARA via the cyclo-oxygenase pathway. EPA is converted through the same pathway into prostaglandin E3, which has 4 to 7- fold less prostaglandin E receptor affinity, is less inflammatory, and may even be pro-apoptotic compared to PGE2. As such, it may be the ratio of ARA to EPA and DHA rather than the absolute levels of marine-derived n-3 PUFAs that contribute most towards their antiproliferative and pro-apoptotic effects.

The ratio of ARA to EPA + DHA can be manipulated through fish oil supplementation, however; genetic factors may play a key role on determining this ratio. Recent genome-wide association and haplotype studies have demonstrated that up to 28% of the additive variance in tissue levels of ARA is explained by variants in a single gene, fatty acid desaturase 1 (FADS1). FADS1 is the rate-limiting enzyme in the conversion of linoleic acid (LA), the most commonly consumed PUFA, to ARA, and homozygotes for the T allele (population frequency of 13%, HapMap -CEU) in rs174537 have lower fatty acid desaturase activity and subsequently lower tissue levels of ARA. While EPA can be produced in vivo from α-linolenic acid, in humans, this process is extremely inefficient and most tissue level EPA derives directly from dietary consumption of fatty fish. Thus, high activity of FAD1 and subsequently increased tissue levels of ARA may offset some of the potential benefits of dietary supplementation with fish oil. To date, no previously published studies have investigated how genetic variants that influence fatty acid desaturase activity might modify the beneficial effects of fish oil supplementation.

The investigators hypothesis is that the individuals with genetically determined lower activity of FADS1 will derive greater benefit from fish oil supplementation than individuals with higher FADS1 activity because of lower tissue levels of ARA and subsequently a more favorable ARA to EPA + DHA ratio. To test this hypothesis the investigators will recruit 150 participants with recently identified adenomatous polyps and conduct a 6-month double blind 3 X 2 factorial randomized controlled trial. The first factor will be the rs174537 genotype (GG, GT, and TT) in the FADS1 gene and the second factor will be fish oil supplementation (fish oil versus placebo). The primary study outcome will be the change from baseline in rectal epithelial cell proliferation as measured by Ki-67 labeling and rectal crypt apoptosis as measured by TUNEL. Secondary endpoints will include rectal epithelial cell expression of COX-2 and 15-PGDH, rectal cell production of PGE2 and PGE3, rectal cell fatty acid concentrations, as well as, changes from baseline in biomarkers of inflammation (C-reactive protein), adipokines (leptin, adiponectin), and markers of insulin sensitivity (HOMA-IR).

The Specific Aims for this research proposal are:

1. to determine the efficacy of fish oil supplements on rectal epithelial cell proliferation indexes and markers of rectal crypt apoptosis; and,
2. to determine the effect of genetically determined fatty acid desaturase activity on fish oil supplementation for markers of colorectal cancer risk.

The investigators long-term objectives are to determine genetic factors that might influence the efficacy of fish oil supplementation in order to conduct a more definitive adenoma recurrence trial using marine-derived n-3 PUFAs. The investigators anticipate that fish oil will have anti-neoplastic effect and individuals with low FADS1 activity will have a greater response compared to individuals with high FADS1 activity. This study will be the first to investigate the nutrigenomics of fish oil supplementation in colorectal cancer chemoprevention and may have implications beyond cancer prevention as fish oil is being actively investigated for its anti-inflammatory effects in cardiovascular and psychiatric diseases as well as diabetes mellitus and the metabolic syndrome.

2. Recruitment and Retention

The investigators will identify eligible participants based on the inclusion criteria by reviewing study data and medical record data collected in the Tennessee Colorectal Polyp Study(TCPS). Participants still eligible after record review will be mailed an introductory letter inviting them to participate. One week after the letter is mailed; a trained interviewer from the Vanderbilt Survey Research Shared Resource (SRSR) will call the potential participants to provide more detailed information about the study, answer questions about the study, and to see if they may be interested in participating. At that time, an appointment will be made with the participant for the baseline in-person visit. After the initial visit and informed consent is obtained an interviewer from the SRSR will conduct the baseline interview survey and 24-hour dietary recalls. At the baseline visit, the investigators will re-genotype rs174535 to confirm the accuracy of the imputation process. This strategy will allow the investigators to efficiently and accurately identify appropriate candidates for our study.

Eligible subjects will present to the Vanderbilt General Clinical Research Center (GCRC) for the initial visit and baseline study procedures. Participants who are eligible for the study and provide written consent for enrollment will have blood obtained; an adipose tissue biopsy performed, and undergoes the baseline rectal mucosal biopsy procedure. Treatment assignment will be obtained from the Vanderbilt Investigational Pharmacy by a coordinator. The first dose of the study medication will be given to patients at the initial visit and the date and time recorded. This date and time will be considered the time of randomization.

3. Randomization

Randomization will be performed according to a permuted block randomization scheme stratified on the three genotypes. Randomization will proceed within these three strata with a block size of balancing interval, varying randomly according to the outcome of a computer generated random number. This ensures that the cumulative proportion of assignments to each treatment will be balanced after each block of assignments has been made.

4. Study Procedures

1. Data Collection

   Because outside dietary exposure to both n-6 and n-3 PUFAs could possibly confound the effect of fish oil supplementation the investigators will perform a total of four 24-hour dietary recall studies for each participant over the course of the study. At enrollment, the investigators will conduct two 24-hour dietary assessments, one on the weekday and one on the weekend, as participants' diet may differ based on the day of the week. In addition the investigators will conduct one 24-hour dietary recall at week 8 and at week 16. The investigators will use data collected from these 24-hour dietary assessments along with standard food composition tables to calculate dietary exposure to PUFAs.

   The investigators will determine adherence to study drug at each in-person visit during the study. Medication and medication changes will be recorded at these visits. Patients who initiate a new NSAID during the study will be withdrawn and an exit visit performed. Adherence to fish oil will also be determined through RBC phospholipid membrane fatty acid analysis performed at month 3 and month 6. In addition, to determine whether fish oil supplementation also influences fatty acid membrane concentration at the target tissue, the investigators will determine the change in rectal epithelial cell phospholipid membrane fatty acid concentration.
2. Fish oil Capsules

   Participants allocated to fish oil supplementation will be instructed to take three Lovaza® capsules each containing 465 mg of EPA and 375 mg DHA daily; this will provide a total daily dose of 1395 mg EPA plus 1125 mg DHA for a total daily dose of fish oil of 2.5 grams. Patients will take one tablet three times a day with meals. Lovaza® capsules are the only FDA approved preparation of fish oil, and as such, the quality of the drug is monitored and assured. Pharmacological grade fish oil capsules have the advantage of providing high concentrations of PUFAs, low levels of contaminants, such as mercury, and almost no fish odor.
3. Placebo Capsules

   The investigators will use oleic acid as a placebo. The reason for the use of oleic acid is several-fold. First, oleic acid (olive oil) capsules have a similar texture, size, color, and consistency to fish oil capsules. More importantly, oleic acid does not undergo conversion to an eicosanoid or any other metabolically active product. This is opposed to corn oil, which has also been used as a placebo in fish oil studies but is primarily linoleic acid and could subsequently increase tissue levels of ARA and confound the results of our study. Oleic acid has been used as a placebo in several prior studies of fish oil supplementation and is well tolerated.
4. Assessment Visits

Patients will attend the GCRC clinic at the baseline (initial visit), after 3 months of study treatment (mid-point visit), and after 6 months of study treatment (end visit). The study coordinator will contact participants every 4 weeks over the course of the study to encourage adherence to the study protocol. At the 3-month and 6-month visits, compliance with treatment will be monitored by capsule count and measurement of RBC phospholipid fatty acid concentrations. Adverse events will be recorded at these visits.

5. Data management and quality control

The Vanderbilt GCRC Informatics Core will be used as a central location for data processing and analysis. Vanderbilt University has developed software tools and workflow methodology for electronic collection and management of research study data. (132) REDCap (Research Electronic Data Capture) is a secure, web-based application that provides an intuitive interface for users to enter validated data remotely (with automated data type and range checks), data manipulation audit trails and reporting, and an export mechanism for end-of-study export of data to common statistical packages.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 and < 80 years of age
* History of 1 or more adenomatous polyps
* Consent to be contacted for future studies
* Participants with known genotype for rs174535 in FADS1
* Prior participation in the Tennessee Colorectal Polyp Study or the Personalized Prevention of Colorectal Cancer Trial

Exclusion Criteria:

* Previously resected colorectal cancer
* Coronary artery disease or congestive heart failure
* Current metabolic or life-threatening disease
* Currently taking fish oil supplements
* Inability or unwillingness to stop NSAIDs or ASA during the study
* Allergic to fish products
* Diagnosis of inflammatory bowel disease
* Diagnosis of any cancer (except non-melanoma skin cancer)
* Diagnosis of liver or kidney disease
* Pregnant or breast feeding

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2018-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey J Murff, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Murff HJ, Shrubsole MJ, Cai Q, Su T, Dooley JH, Cai SS, Zheng W, Dai Q. N-3 Long Chain Fatty Acids Supplementation, Fatty Acids Desaturase Activity, and Colorectal Cancer Risk: A Randomized Controlled Trial. Nutr Cancer. 2022;74(4):1388-1398. doi: 10.1080/01635581.2021.1955286. Epub 2021 Jul 22. PMID 34291724

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Started | 26 | 25 | 25 | 26 | 19 | 20
Completed | 24 | 20 | 22 | 24 | 16 | 18
Not Completed | 2 | 5 | 3 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo | Total
Number analyzed (Participants) | 26 | 25 | 25 | 26 | 19 | 20 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.7) | 60 (8.3) | 59.6 (9.6) | 58.9 (7.4) | 60.5 (9.8) | 61.6 (7.6) | 59.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 7 | 12 | 8 | 8 | 68
  Male | 7 | 11 | 18 | 14 | 11 | 12 | 73

OUTCOME MEASURES:

1. Primary Outcome: Rectal Epithelial Cell Proliferation
Description: The primary outcome of interest is rectal epithelial cell proliferation, as measured by Ki67 (mib-1) labeling. Expression of Ki-67 in colon epithelial cells will be detected following the standard IHC protocol of EnVision™+ System, HRP (DAKO).
Time Frame: 6 month
Population: Patients with before and after rectal biopsies
Measure: Mean (Standard Deviation); unit: percentage of cells positive
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
percentage of cells positive | 19.3 (6.8) | 20.3 (7.6) | 18.9 (8.5) | 16.8 (6.2) | 15.7 (5.4) | 20.8 (6.7)

2. Primary Outcome: Rectal Epithelial Cell Apoptosis
Description: The primary outcome of interest is rectal epithelial cell apoptosis as measured by TUNEL (TdT-mediated dUTP Nick-End Labeling). The TUNEL assay is conducted to measure apoptosis of colon epithelium using DeadEnd Colorimetric TUNEL System (Promega). After all fields of each sample are measured, the final immunoreaction indices are generated automatically by setting algorithms as ''total positive area / total nuclear area. Apoptotic activity is also scored using standard morphologic criteria applied to H&E stained sections.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of cells positive
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
percentage of cells positive | 1.17 (1.79) | 1.30 (1.30) | 1.00 (1.27) | 2.61 (4.55) | 1.44 (1.77) | 1.33 (1.78)

3. Secondary Outcome: Rectal Epithelial Cell COX-2 Expression
Description: Expression of COX-2 in rectal epithelial cells will be detected following the standard IHC protocol of EnVision™+ System, HRP (DAKO).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of cells positive
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
percentage of cells positive | 6.47 (4.40) | 4.62 (2.81) | 5.10 (3.05) | 5.31 (3.32) | 2.86 (1.40) | 5.86 (4.29)

4. Secondary Outcome: Rectal Epithelial Cell 15-PGDH Expression
Description: Expression of 15-PGDH in rectal epithelial cells will be detected following the standard IHC protocol of EnVision™+ System, HRP (DAKO).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of cells positive
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
percentage of cells positive | 27.5 (8.14) | 27.6 (4.58) | 25.1 (6.42) | 29.3 (6.3) | 23.8 (8.5) | 27.1 (6.15)

5. Secondary Outcome: Rectal Epithelial Cell Phospholipid Fatty Acid Content
Description: Lipids will be extracted using the method of Folch-Lees
Time Frame: 6 months
Population: Due to inadequate rectal tissue specimens we were unable to measure rectal tissue phospholipids
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Rectal Epithelial Cell Production of PGE2 and PGE3
Description: liquid chromatography/tandem mass spectrometric on rectal biopsy samples
Time Frame: 6 months
Population: For some participants the volume of frozen tissue was not enough to measure rectal eicosanoids and are not included in the analysis (2 from GG, fish oil, 2 from GG, placebo, 3 from GT fish oil, 4 GT placebo, 1 TT fish oil and 3 TT placebo)
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 22 | 18 | 19 | 20 | 15 | 15
ng/g
  PGE2 | 11.4 (13.3) | 23.6 (33.4) | 14.4 (19.7) | 22.1 (40.0) | 16.6 (14.1) | 24.4 (27.7)
  PGE3 | 1.40 (1.87) | 2.89 (3.38) | 2.10 (2.00) | 2.63 (2.98) | 4.43 (9.04) | 1.84 (2.00)

7. Other Pre Specified Outcome: C-reactive Protein
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
mg/L | 3.98 (6.64) | 3.87 (7.13) | 2.11 (2.23) | 4.96 (6.92) | 2.58 (4.00) | 2.34 (2.85)

8. Other Pre Specified Outcome: Adipokines
Description: leptin and adiponectin
Time Frame: 6 months
Population: Adipokines were not measured on all trial participants due to assay expense. Samples measurements were not completed on 3 GG, fish oil, 0 GG, placebo, 3 GT fish oil, 4 GT placebo, 7 TT fish oil, 9 TT placebo
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 21 | 20 | 19 | 20 | 9 | 9
ng/mL
  Leptin | 25.3 (19.0) | 24.0 (30.1) | 20.2 (15.7) | 27.9 (22.0) | 10.9 (8.62) | 23.0 (26.4)
  Adiponectin | 22.4 (25.8) | 20.5 (17.9) | 18.9 (13.4) | 14.9 (13.9) | 29.4 (33.9) | 15.3 (7.03)

9. Other Pre Specified Outcome: Insulin Sensitivity
Description: homeostasis model assessment-insulin resistance (HOMA-IR) HOMA-IR. Fasting insulin and glucose were be used to determine HOMA-IR: [fasting glucose (mmol/l) x fasting insulin (µU/ml)]/22.5]", Optimal insulin sensitivity: < 1, Early insulin resistance: > 1.9, Significant insulin resistance: > 2.9
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: HOMA-IR Index
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
Number analyzed (Participants) | 24 | 20 | 22 | 24 | 16 | 18
HOMA-IR Index | 0.67 (0.56) | 0.98 (0.92) | 0.67 (0.57) | 1.01 (1.33) | 0.72 (0.75) | 0.80 (0.75)

ADVERSE EVENTS:
Time Frame: 6 months
Description: For the purposes of this study and adverse event is defined as any untoward medical occurrence in a subject, not necessarily having a causal relationship with the study. A serious adverse event (SAE) is any untoward medical occurrence that a) results in death, b) is life-threatening, c) requires inpatient hospitalization or prolongation of existing hospitalization, d) results in persistent or significant disability/incapacity, or e) is a congenital anomaly/birth defect.
Arm/Group | rs174535 (GG), Fish Oil Supplements | rs174535 (GG), Placebo | rs174535 (GT), Fish Oil Supplements | rs174535 (GT), Placebo | rs174535 (TT), Fish Oil Supplement | rs174535 (TT), Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/26 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/25 | 0/25 | 0/26 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 1/26 | 0/25 | 0/25 | 0/26 | 2/19 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rs174535 (GG), Fish Oil Supplements (N=26) | rs174535 (GG), Placebo (N=25) | rs174535 (GT), Fish Oil Supplements (N=25) | rs174535 (GT), Placebo (N=26) | rs174535 (TT), Fish Oil Supplement (N=19) | rs174535 (TT), Placebo (N=20)
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Study subject presented to emergency room with chest pain. The subject was admitted and diagnosed with a myocardial infarction. This was a serious adverse events but deemed not related to study participation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rs174535 (GG), Fish Oil Supplements (N=26) | rs174535 (GG), Placebo (N=25) | rs174535 (GT), Fish Oil Supplements (N=25) | rs174535 (GT), Placebo (N=26) | rs174535 (TT), Fish Oil Supplement (N=19) | rs174535 (TT), Placebo (N=20)
Bloating and eructations (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Unable to tolerate the medication due to gastrointestinal side effects involving bloating and eructations

LIMITATIONS AND CAVEATS:
Did not reach target accrual rate in T/T arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT01661764/Prot_SAP_000.pdf